CLINICAL TRIAL: NCT02314819
Title: A Randomized, Double-blind and Placebo-controlled Phase III Trial Comparing Fruquintinib Efficacy and Safety vs Best Support Care (BSC) in Advanced Colorectal Cancer Patients Who Have Failed at Least Second Lines of Chemotherapies
Brief Title: A Phase III Trial Evaluating Fruquintinib Efficacy and Safety in 3+ Line Colorectal Cancer Patients （FRESCO)
Acronym: FRESCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Fudan University (Other); Eighty-One Hospital of People's Liberation Army (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-013-00CH1
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment arm (Active Comparator): treatment arm- subjects will receive Fruquintinib 5mg orally, QD, plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Interventions: Drug: fruquintinib
- control arm (Placebo Comparator): control arm- subjects will receive Fruquintinib placebo 5mg orally, QD, plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fruquintinib — fruquintinib is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
  Other Names: HMPL-013
  Arms: treatment arm
Drug: placebo — fruquintinib placebo is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
  Other Names: HMPL-013 placebo
  Arms: control arm

SUMMARY:
Fruquintinib administered at 5mg once daily(QD) in 4 weeks treatment cycle (three weeks on and one week off) was well tolerated and demonstrated encouraging preliminary clinical antitumor activity in patients with metastatic colorectal cancer (CRC) in phase Ib and phase 2 study. This study is aimed to evaluate the efficacy and safety of Fruquintinib in the treatment of patients with metastatic CRC who have progressed after second line or above standard chemotherapy

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter Phase III clinical trial to compare the efficacy and safety of Fruquintinib plus BSC versus placebo plus BSC in patients with metastatic colorectal cancer who have progressed after second-line or above standard chemotherapy. After checking eligibility criteria, subjects will be randomized into Fruquintinib plus BSC group (treatment group) or placebo plus BSC group (control group) in a ration of 2:1. Primary Efficacy Endpoint: Overall Survival (OS). Secondary Efficacy Endpoints: Progression free survival (PFS) (According to RECIST Version 1.1), Objective Response Rate (ORR), Disease Control Rate (DCR), . Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age , with ≥ 40Kg
* Histological or cytological confirmed colorectal cancer
* ECOG performance status of 0-1
* Standard regimen failed or no standard regimen available
* Adequate hepatic, renal, heart, and hematologic functions
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure

Exclusion Criteria:

* - Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Evidence of CNS metastasis
* Intercurrence with one of the following: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial - Previous treatment with VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Proteinuria ≥ 2+ (1.0g/24hr)
* Have evidence or a history of bleeding tendency within two months of the enrollment, regardless of seriousness
* Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Within 6 months before the first treatment occurs acute myocardial infarction, acute coronary syndrome or CABG
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
overall survival | from randomization until death due to any cause, assessed up to 2 year
  every two months after end of treatment (EOT) observation period at 30 days after the last medication

SECONDARY OUTCOMES:
progression free survival | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Objective Response Rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease Control Rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to within 30 days after the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, MD, Principal Investigator — Fudan University
Locations (15):
- China (15):
  - Hutchison Medi Pharma Investigational Site, Hefei, Anhui
  - Hutchison Medi pharma Investigational Site, Beijing, Beijing Municipality
  - Hutchison Medi Pharma Investigational Site, Guangzhou, Guangdong
  - Hutchison Medi Pharma investigational site, Shenzhen, Guangdong
  - Hutchison Medi Pharma Investigational Site, Liuchow, Guangxi
  - Hutchison Medi Pharma Investigational Site, Harbin, Heilongjiang
  - Hutchison Medi Pharma Investigational Site, Changsha, Hunan
  - Hutchison Medi Pharma Investigational Site, Changzhou, Jiangsu
  - Hutchison Medi Pharma Investigational Site, Nanjing, Jiangsu
  - Hutchison Medi Pharma Investigational Site, Nantong, Jiangsu
  - Hutchison Medi Pharma Investigational Site, Xuzhou, Jiangsu
  - Hutchison Medi Pharma Investigational Site, Changchun, Jilin
  - Hutchison Medi Pharma Investigational Site, Qingdao, Shandong
  - Hutchison Medi Pharma Investigational Site, Shanghai, Shanghai Municipality
  - Hutchison Medi Pharma Investigational Site, Hangzhou, Zhejiang

REFERENCES:
- [Result] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Derived] Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Wang N, Zhang B, Zhang Q, Su W, Guo X, Li J. Subgroup Analysis by Liver Metastasis in the FRESCO Trial Comparing Fruquintinib versus Placebo Plus Best Supportive Care in Chinese Patients with Metastatic Colorectal Cancer. Onco Targets Ther. 2021 Aug 11;14:4439-4450. doi: 10.2147/OTT.S307273. eCollection 2021. PMID 34408440
- [Derived] Xu R, Qin S, Guo W, Bai Y, Deng Y, Yang L, Chen Z, Zhong H, Pan H, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Xu J, Chen D, Li W, Sun S, Yu Z, Cao P, Li J, Chen H, Wang J, Wang S, Wang H, Wang N, Zhang B, Han R, Su W, Guo X, Li J. Subgroup analysis by prior anti-VEGF or anti-EGFR target therapy in FRESCO, a randomized, double-blind, Phase III trial. Future Oncol. 2021 Apr;17(11):1339-1350. doi: 10.2217/fon-2020-0875. Epub 2020 Dec 16. PMID 33325251
- [Derived] Li J, Guo W, Bai Y, Deng Y, Yang L, Chen Z, Zhong H, Xu R, Pan H, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Xu J, Chen D, Li W, Sun S, Yu Z, Cao P, Shen L, Chen H, Wang S, Wang H, Fan S, Guo X, Wang N, Han R, Zhang B, Qin S. Safety Profile and Adverse Events of Special Interest for Fruquintinib in Chinese Patients with Previously Treated Metastatic Colorectal Cancer: Analysis of the Phase 3 FRESCO Trial. Adv Ther. 2020 Nov;37(11):4585-4598. doi: 10.1007/s12325-020-01477-w. Epub 2020 Sep 8. PMID 32901330